CLINICAL TRIAL: NCT02881866
Title: Specificity of Dyspnoea Relief With Inhaled Furosemide
Acronym: FurosAH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Joanna Grogono, Clinical Research Fellow, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UREC150939
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Dyspnea
Keywords: Air hunger; Work/effort; Aerosolized; Hypercapnia; Resistive load; Nebulised
MeSH Terms: conditions — Dyspnea; Hypercapnia | interventions — Furosemide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Hunger (Active Comparator): Previous studies have shown that inhaled furosemide relieves 'air hunger'.
  Each volunteer has 3 mists per visit. The mists are either in the order of Furosemide-Saline-Furosemide or Saline-Furosemide-Saline. The furosemide mist is 40mg (10mg/ml) nebulised and the saline mist is 4ml nebulised.
  Induced air hunger (hypercapnia with constrained ventilation) is the active comparator and will be the type of breathlessness induced, before and after each mist inhalation on one day. .
  Interventions: Drug: Furosemide; Drug: Saline
- Work Effort (Experimental): Induced sense of breathing effort (raised ventilation with external resistive load) is the 'experimental arm' and will be the type of breathlessness induced, before and after each mist inhalation on the other day. .
  Interventions: Drug: Furosemide; Drug: Saline

INTERVENTIONS:
Drug: Furosemide
  Other Names: Lasix
Drug: Saline
  Other Names: 0.9% sodium chloride

SUMMARY:
This study evaluates the effect of inhaled furosemide on different types of breathlessness relief in healthy volunteers. Each volunteer inhaled mists of either furosemide or a control substance on 3 occasions per day on 2 separate days. On one day they performed one breathlessness test which creates an 'urge to breathe' known as air hunger (AH) and the other day they performed a breathlessness test which increases the sense of work/effort (WE) of breathing. The study is double blinded so neither the volunteer or the research knows which mist is being inhaled.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled trial. 16 healthy volunteers will attend 4 sessions. After 2 practice sessions subjects will undergo 2 test days where they will be made to feel 'air hunger' (hypercapnia with constrained ventilation) before and after mist inhalations on one day and sense of breathing 'effort' (raised ventilation with external resistive load) before and after mist inhalations on the second test day. The mist will either be furosemide or a placebo (saline) mist.

The urge to urinate from systemic absorption from the lungs will be accounted for by a concomitant administration of intravenous furosemide when saline is inhaled.

Furosemide is a prescription drug which makes kidneys produce more urine. When administered by inhalation as an aerosol it has direct action in the lungs which sensitises slowly adapting stretch receptors which is believed to account for the relief of dyspnoea previously reported with inhaled furosemide.

Vagal afferents from the pulmonary stretch receptors are known to be involved in relief of air hunger but it is not known if they will also relieve the sense of breathing effort. Relief of breathlessness will be measured and compared between the two trial days to see if furosemide specifically relieves the 'air hunger' type of breathlessness and not the 'effort' type of breathlessness.

ELIGIBILITY:
Inclusion Criteria:

- Healthy individuals

Exclusion Criteria:

* On any medication, including herbal medication (other than mild analgesics, vitamins and mineral supplements or, for females, oral contraceptives), whether prescribed or over-the-counter, in the two weeks prior to test sessions involving administration of furosemide or saline.
* Female participants who are pregnant, lactating or planning pregnancy over the course of trial
* A medical history of heart, kidney or liver disease/electrolyte disturbances/ immunosuppression/frequent fainting episodes/COPD/nasal polyps/Addison's/acute porphyria/significant prostatic symptoms/acute gout attack/life expectancy <6months or history of allergic reaction to furosemide and/or any of the other ingredients of furosemide or amiloride, sulfonamides or sulphonamide derivatives, such as sulfadiazine or co-trimoxazole
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Have participated in another research trial involving an investigational product in the past 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale for breathlessness type | 20minutes
  The visual analogue scale (VAS) is from 0 (no breathlessness) to 100 (maximal breathlessness willing to tolerate). The VAS is measure every 15-20 seconds during each experimentally induced breathing test. Each breathing test is performed before and after each mist inhalation. Total of 6 breathing tests. The final minute of a 4 minute steady state breathing test is analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna C Grogono, MBBS, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moosavi SH, Binks AP, Lansing RW, Topulos GP, Banzett RB, Schwartzstein RM. Effect of inhaled furosemide on air hunger induced in healthy humans. Respir Physiol Neurobiol. 2007 Apr 16;156(1):1-8. doi: 10.1016/j.resp.2006.07.004. Epub 2006 Aug 28. PMID 16935035
- [Background] Nishino T, Ide T, Sudo T, Sato J. Inhaled furosemide greatly alleviates the sensation of experimentally induced dyspnea. Am J Respir Crit Care Med. 2000 Jun;161(6):1963-7. doi: 10.1164/ajrccm.161.6.9910009. PMID 10852774
- [Derived] Grogono JC, Butler C, Izadi H, Moosavi SH. Inhaled furosemide for relief of air hunger versus sense of breathing effort: a randomized controlled trial. Respir Res. 2018 Sep 20;19(1):181. doi: 10.1186/s12931-018-0886-9. PMID 30236110